CLINICAL TRIAL: NCT04875143
Title: Effects Of Acute Supplementation Of Citrus Aurantium L. On The Recovery Of Autonomic And Cardiovascular Activity After A Submitted Aerobic Exercise Session In Healthy Individuals: A Prospective, Randomizado-Plato-Rudomizado Plado Study.
Brief Title: Effects Of Acute Supplementation Of Citrus Aurantium L. On The Recovery Of Autonomic And Cardiovascular Activity After A Sub-Maximum Aerobic Exercise Session In Healthy Individuals
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pernambuco (Other)
Responsible Party: Principal Investigator, Cicero Jonas R Benjamim, Student, University of Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: x32
Record Dates: First submitted 2021-04-30; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: To Evaluate the Effect of Supplementation of Citrus Aurantium in Active Individuals

STUDY DESIGN:
Intervention Model Description: One hour before the experimental procedures, the volunteers will ingest 500 mg of Citrus aurantium L. extract or starch (placebo) in capsules according to the selected protocol. Neither the researcher nor the volunteer will know if the capsule is a placebo or Citrus aurantium L. (double-blind and placebo-controlled) Before starting these protocols, a heart rate monitor (Polar RS800CX, Finland) will be placed on the volunteers to record the HR beat to beat during the entire collection. After ingestion of the capsules, the volunteers will remain in initial rest sitting for 15 minutes. During rest, HR, systolic blood pressure (SBP), diastolic blood pressure (DBP) and respiratory rate (RF) values will be recorded in the 15th minute.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: From a pre-established randomization, on the first day of collection, volunteers will be allocated to group I (Placebo) or group II (Citrus aurantium L.). In the first intervention, the volunteers allocated to group I will take a capsule containing 500mg of starch, at the end of this, another capsule containing 500mg of Citrus aurantium L. will be provided for the second intervention. Conversely, the volunteers allocated to group II will ingest a capsule containing 500mg of Citrus aurantium L. in the first intervention, and at the end of the experiment, another capsule containing 500mg of starch will be provided.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PLACEBO (Placebo Comparator): From a pre-established randomization, on the first day of collection, volunteers will be allocated to group I (Placebo) or group II (Citrus aurantium L.). In the first intervention, the volunteers allocated to group I will take a capsule containing 500mg of starch, at the end of this, another capsule containing 500mg of Citrus aurantium L. will be provided for the second intervention. Conversely, the volunteers allocated to group II will ingest a capsule containing 500mg of Citrus aurantium L. in the first intervention, and at the end of the experiment, another capsule containing 500mg of starch will be provided.
  Interventions: Dietary Supplement: Citrus aurantium L.
- Citrus aurantium L. (Experimental): From a pre-established randomization, on the first day of collection, volunteers will be allocated to group I (Placebo) or group II (Citrus aurantium L.). In the first intervention, the volunteers allocated to group I will take a capsule containing 500mg of starch, at the end of this, another capsule containing 500mg of Citrus aurantium L. will be provided for the second intervention. Conversely, the volunteers allocated to group II will ingest a capsule containing 500mg of Citrus aurantium L. in the first intervention, and at the end of the experiment, another capsule containing 500mg of starch will be provided.
  Interventions: Dietary Supplement: Citrus aurantium L.

INTERVENTIONS:
Dietary Supplement: Citrus aurantium L. — In the first intervention, the volunteers allocated to group I will take a capsule containing 500mg of starch, at the end of this, another capsule containing 500mg of Citrus aurantium L. will be provided for the second intervention.
  Other Names: Sour orange

SUMMARY:
INTRODUCTION: Non-pharmacological interventions for the treatment of cardiovascular and metabolic disorders have been investigated. In this context, Citrus aurantium L., popularly known as Bitter Orange, rich in synephrine (p-synephrine), a phenylethylaminic alkaloid that is present in the bitter orange peel, has been used as an adjunct in metabolic disorders. Given the effects, the components of Citrus aurantium L. diverge from other thermogens by being able to activate metabolism and lipolysis without interfering with the performance of the cardiovascular system, making this an advantage for its use in diets. In studies, it has been observed that the activation of β-3 receptors plays an important role in the regulation and activation of other receptors, modulating and, when they are stimulated in excess, and thus, it presents effects that in addition to not causing overload in the cardiovascular system. OBJECTIVE: To evaluate the effect of supplementation of Citrus aurantium L. in combination with submaximal aerobic exercise on autonomic and cardiovascular parameters of physically active. METHODOLOGY: This is a prospective, randomized, placebo-controlled, double-blind crossover trial. 40 physically active volunteers will participate in the study. They will be qualified for the voluntary study of the male gender, who are aged between 18 and 30 years old and have a Body Mass Index (BMI) between 18.5 kg / m² and 29.9 kg / m². Do not use any medication that may interfere with cardiac autonomic modulation and do not have skeletal muscle damage. They will be considered as exclusion criteria for clinical patients, as well as those who have already used anabolic steroids or who have cardiorespiratory, neurological disorders and other known impairments that prevent the subject from performing the procedures. EXPECTED RESULTS: Speculated that the protective effects of flavonoids and their antioxidant properties found in Citrus aurantium L., optimize autonomic recovery after aerobic exercise. In addition, HRV can be used to ascertain its SNA activation effects and validate the safety of the applicability of this supplement for overweight populations, considering that it is used for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers, aged between 18 and 30 years and with a Body Mass Index (BMI) between 18.5 kg / m² and 29.9 kg / m² will be considered eligible for the study.

Exclusion Criteria:

* Smoking patients will be considered as exclusion criteria. As well as individuals with cardiorespiratory, neurological disorders and other known impairments that prevent the subject from performing the procedures.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | through study completion, an average of 1 year
  Heart rate variability (HRV) is a non-invasive method that analyzes the autonomic regulation of heart rate in humans. It is a conventionally accepted term to describe oscillations in the intervals between consecutive heartbeats (RR intervals), which are related to the influences of the ANS on the sinus node. It is a non-invasive technique, whose analysis can be performed using linear methods, in the domain of time and frequency, and non-linear, in the domain of chaos

SECONDARY OUTCOMES:
Blood pressure | through study completion, an average of 1 year
  Check the blood pressure of subjects with and without the ingestion of Citrus aurantium L. before and in the recovery period after physical exercise;

CONTACTS AND LOCATIONS:
Locations (1):
- Cicero Jonas Rodrigues Benjamim, Juazeiro do Norte, Ceará, Brazil